CLINICAL TRIAL: NCT05693493
Title: Can Proprioceptive Knee Brace Improve Functional Outcome Following Total Knee Arthroplasty?
Brief Title: Can Proprioceptive Knee Brace Improve Functional Outcome Following TKA?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022.223-T
Record Dates: First submitted 2022-12-14; First posted 2023-01-23 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee brace; Knee OA; Proprioceptive knee brace; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Device: Proprioceptive knee brace Subjects will use proprioceptive knee brace for 6 weeks post-op, in addition to basic management such as physiotherapy.
  Interventions: Device: Proprioceptive knee brace
- Control group (No Intervention): No device. Subjects will receive basic management such as physiotherapy.

INTERVENTIONS:
Device: Proprioceptive knee brace — For the intervention group that randomly consisted of 15 subjects will be using a design of knee brace (Reaction Web®; DonJoy, Vista, CA). The elastomeric web design helps to reduce pain by dispersing load across the knee. The web acts like a spring to absorb shock and shifts the peak loads away from the painful area of the knee. Elastomeric web acts to dynamically stabilise the patella on all sides, bringing the patella into proper tracking position to reduce pain for patients with general patellofemoral instabilities. Reaction Web® has dual-axis hinges that are flexible, creating synergy with the elastomeric web for optimal fit and support, and providing energy dispersion to the knee.
  Arms: Intervention group

SUMMARY:
Osteoarthritis is among the most prevalent form of degenerative joint disease in arthritis. The World Health Organisation identified osteoarthritis as one of the top ten most disabling cause of disease in developed countries, and the single most common cause of disability for elderly persons. In fact, worldwide statistics for men and women over 60 years of age with signs of symptomatic osteoarthritis are estimated to be at 9.6% and 18.0% respectively. In Hong Kong, the latest census revealed that 514,000 people suffer from degenerative arthritis, representing 0.7% of the population. Although these values are much lower than the international figures reported by the WHO, it is inevitable that the prevalence of osteoarthritis will continue to rise with an increasing trend of obesity and an aging population in Hong Kong. Similar to any other chronic disease with wide prevalence, the impact of osteoarthritis translates to a substantial socioeconomic burden on a societal level.

Total knee arthroplasty has become the gold standard to manage the pain and disability associated with end-stage arthritis who have exhausted all conservative measures. Although contemporary advances in prosthesis design, surgical techniques, postoperative rehabilitation regimes have hasten patient's recovery, the restoration of proprioception and neuromuscular control is often prolonged despite solid rehabilitation regimes.

Knee bracing is one of the non-pharmacological modalities designed to evenly distribute load and provide proprioceptive feedbacks for those with knee injuries or knee pain. There are four categories of knee braces for the purpose of prophylactic, functional, rehabilitative and unloader/off-load. This study will mainly be focusing on the effects of the unloader/off-loader brace. Previous studies have demonstrated the effects on alteration of kinematic variables, including range of movement (p=0.002), speed of walking (p<0.001) and knee adduction moment (p=0.001) for knee injuries and osteoarthritis as a part of the conservative management protocol. However, there have few studies that investigated whether proprioceptive knee bracing has any role in functional recovery post total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age over 18 years old) underwent Total Knee Arthroplasty within 2 to 4 weeks;
2. Adult who is able to provide written consent and compliance with treatment and assessment regime

Exclusion Criteria:

1. Patients with disabilities, wheelchair dependence for mobility;
2. Underwent revision Total Knee Arthroplasty;
3. Found with complication wounds following surgery;
4. Diagnosed with comorbidities e.g. inflammatory arthritis, obesity, dermatological disorders that might affect their compliance to treatment;
5. Do not fit to the sizes of knee braces;
6. Not to given written consent and be non-compliance with the treatment and assessment regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes of the time of 6-meter test | pre-op, 6-weeks, 6-months and 12-months post-op
  The 6-meter test timed walking gait test has been documented to be a valid and reliable substitute. Patients will be asked to walk a straight line of 6 meters where the time taken to complete the distance will be measured. (<7.5 seconds is normal).
Changes of the time of Time up and go test (TUG) | pre-op, 6-weeks, 6-months and 12-months post-op
  The Time up and go test (TUG) is to determine fall risk and measure the progress of balance, sit to stand and walking. Patients will be asked to stand up from a chair, walk as quickly as possible in their a safe and most comfortable gait until they pass to 3 meters (10 feet) end of marked course with both feet. Turn around and walk back to the chair, time will be counted to the moment until the back of patients touches the back of the chair.
Change in the range of motion | pre-op, 6-weeks, 6-months and 12-months post-op
  The active range of motion test predicts the mobility of the joint by measuring the amount of active knee extension and flexion. Knee extension: The patient is supine. The heel of the limb of interest is propped on a bolster, assuring the back of the knee and calf are not touching the support surface. The patient is asked to actively contract the quadriceps. The amount of knee extension is recorded with the goniometer. Knee flexion: The patient is prone. The patient flexes the knee as far as possible. The amount of knee flexion is recorded with the goniometer."

SECONDARY OUTCOMES:
Knee extensor/flexor strength | pre-op, 6-weeks, 6-months and 12-months post-op
  Muscle strength on the quadriceps is measured by instructing the patient to perform an active knee extension movement in a sitting position with both feet free from ground, and the hip and knee joint flexed at 90%. The optimal isometric force of the knee extension/flexion movement is measured by the dynamometer attached at the malleoli level with a strap.
  The measurements will be taken at maximum force for three times.
Short-form 12 | pre-op, 6-weeks, 6-months and 12-months post-op
  The SF-12 health survey uses 12 questions to measure patient's functional health and well-being from a patient's point of view. It is reliable and validated measure that summaries the patients' physical and mental health. The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | pre-op, 6-weeks, 6-months and 12-months post-op
  The WOMAC questionnaire is a questionnaire that measures patient's pain, stiffness and physical function and can be summed up into a score out of 96. A high score indicates a more disabled participant.
The Forgotten Joint Score-12 | pre-op, 6-weeks, 6-months and 12-months post-op
  The FJS-12 comprise measures for the assessment of joint-specific patient-reported outcome in their ability to forget about a joint as a result of successful treatment. Join awareness can be simply defined as any unintended perception of a joint.
  It is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities
Knee stability test | pre-op, 6-weeks, 6-months and 12-months post-op
  KT-1000 will be used at the assessing of knee laxity as it provides an objective evaluation of knee stability resulting from the automated anterior drawer test it performs.
Knee Society Score (KSS) | pre-op, 6-weeks, 6-months and 12-months post-op
  The KSS is an instrument assessing patient's pain and functionality based on a series of questions interviewed by a clinician. The validated questionnaire combines the objective physician derived component with a subjective patient derived component which evaluates pain, functionality, satisfaction and fulfillment of expectations. The results will be calculating the total score with 100 being the highest and 0 the lowest.
Knee Society Function Score (KFS) | pre-op, 6-weeks, 6-months and 12-months post-op
  The validated questionnaire combines the objective physician derived component with a subjective patient derived component which evaluates pain, functionality, satisfaction and fulfillment of expectations. The results will be calculating the total score with 100 being the highest and 0 the lowest.
Clinical Research Compliance assessment: compliance to intervention | 6-weeks, 6-months and 12-months post-op
  Clinical Research Compliance assessment will be conducted to measures the period and amount of time designated knee brace has been put on as interventional means.
Clinical Research Compliance assessment: compliance to routine physiotherapy | 6-weeks, 6-months and 12-months post-op
  It recorded the attendance of routine post-operative procedures of physiotherapy training one might receive.
Patients satisfaction Survey | pre-op, 6-weeks, 6-months and 12-months post-op
  Patients satisfaction Survey is to be recorded in terms not only how well to the quality of care patient was being treated, but to also the content a patient is with the care they received.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tim-Yun Ong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers

DOCUMENTS (2):
  • Study Protocol (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT05693493/Prot_000.pdf
  • Informed Consent Form (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT05693493/ICF_001.pdf